CLINICAL TRIAL: NCT03383458
Title: A Phase 3, Randomized, Double-blind Study of Adjuvant Nivolumab Versus Placebo for Participants With Hepatocellular Carcinoma Who Are at High Risk of Recurrence After Curative Hepatic Resection or Ablation
Brief Title: A Study of Nivolumab in Participants With Hepatocellular Carcinoma Who Are at High Risk of Recurrence After Curative Hepatic Resection or Ablation
Acronym: CheckMate 9DX
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-9DX
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2017-12-21; First posted 2017-12-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Biological: Nivolumab
- Arm B (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Arm A
Other: Placebo — specified dose on specified days
  Arms: Arm B

SUMMARY:
This study will investigate if nivolumab will improve recurrence-free survival (RFS) compared to placebo in participants with HCC who have undergone complete resection or have achieved a complete response after local ablation, and who are at high risk of recurrence

ELIGIBILITY:
Inclusion Criteria:

* Participants with a first diagnosis of HCC who have undergone a curative resection or ablation
* Participants are eligible to enroll if they have non-viral related-HCC, or if they have HBV-HCC, or HCV-HCC
* Child-Pugh Score 5 or 6
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Any evidence of tumor metastasis or co-existing malignant disease
* Participants previously receiving any prior therapy for HCC, including loco-regional therapies
* Participants who have undergone a liver transplant or those who are in the waiting list for liver transplantation
* Participants who have received a live/attenuated vaccine within 30 days of randomization (eg, varicella, zoster, yellow fever, rotavirus, oral polio and measles, mumps, rubella [MMR]).

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2031-02-27 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free Survival (RFS) | Up to 49 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 7 years
Time to recurrence (TTR) | Up to 49 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (184):
- United States (28):
  - Local Institution - 0081, Anniston, Alabama
  - Mayo Clinic in Arizona - Phoenix, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Local Institution - 0135, Los Angeles, California
  - Local Institution - 0088, Palo Alto, California
  - Local Institution - 0085, San Francisco, California
  - Local Institution - 0235, Aurora, Colorado
  - Local Institution - 0267, Miami, Florida
  - Sylvester Comprehensive Cancer Center/ UMHC, Miami, Florida
  - Local Institution - 0163, Tampa, Florida
  - Local Institution - 0009, Atlanta, Georgia
  - Local Institution - 0025, Westwood, Kansas
  - Local Institution - 0086, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Local Institution - 0209, St Louis, Missouri
  - Local Institution - 0075, New York, New York
  - Local Institution - 0208, New York, New York
  - Local Institution - 0045, New York, New York
  - Local Institution - 0219, White Plains, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - Local Institution - 0206, Portland, Oregon
  - Local Institution - 0272, Austin, Texas
  - Local Institution - 0270, Dallas, Texas
  - Local Institution - 0156, Dallas, Texas
  - Local Institution - 0273, Tyler, Texas
  - McGuire VA Medical Center, Richmond, Virginia
  - Local Institution - 0154, Seattle, Washington
- Argentina (3):
  - Local Institution - 0243, Gorriti, Buenos Aires
  - Local Institution - 0254, Pilar, Buenos Aires
  - Local Institution - 0244, Rosario, Santa Fe Province
- Australia (7):
  - Local Institution - 0239, Blacktown, New South Wales
  - Local Institution - 0166, Camperdown, New South Wales
  - Local Institution - 0141, Concord, New South Wales
  - Local Institution - 0220, Herston, Queensland
  - Local Institution - 0164, Adelaide, South Australia
  - Local Institution - 0224, Heidelberg, Victoria
  - Local Institution - 0124, Nedlands, Western Australia
- Austria (3):
  - Local Institution - 0012, Graz
  - Local Institution - 0003, Vienna
  - Local Institution - 0001, Vienna
- Belgium (5):
  - Local Institution - 0033, Brussels
  - Local Institution - 0064, Brussels
  - Local Institution - 0068, Edegem
  - Local Institution - 0071, Ghent
  - Local Institution - 0108, Leuven
- Brazil (7):
  - Local Institution - 0090, Belo Horizonte, Minas Gerais
  - Local Institution - 0275, Barretos, São Paulo
  - Local Institution - 0237, Cerqueira César, São Paulo
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, São Paulo, São Paulo
  - Local Institution - 0023, São Paulo
  - Local Institution - 0236, São Paulo
- Canada (2):
  - Local Institution, Calgary, Alberta
  - Local Institution - 0116, Edmonton
- Chile (4):
  - Local Institution - 0247, Viña del Mar, Región de Valparaíso
  - Local Institution - 0248, Santiago, Santiago Metropolitan
  - Local Institution - 0246, Santiago, Santiago Metropolitan
  - Local Institution - 0245, Santiago, Santiago Metropolitan
- Local Institution - 0256, Bogotá, Colombia
- France (16):
  - Local Institution - 0057, Bobigny
  - Local Institution - 0052, Brest
  - CHU Estaing, Clermont-Ferrand
  - Local Institution - 0046, Clichy
  - Local Institution - 0061, Créteil
  - Local Institution - 0013, Grenoble
  - Local Institution - 0222, Lille
  - Local Institution - 0051, Lyon
  - Local Institution - 0043, Montpellier
  - Local Institution - 0037, Nice
  - Local Institution, Poitiers
  - Local Institution - 0098, Reims
  - Local Institution - 0212, Rennes
  - Local Institution - 0044, Saint-Priest-en-Jarez
  - Local Institution - 0011, Vandœuvre-lès-Nancy
  - Local Institution - 0054, Villejuif
- Germany (15):
  - Local Institution - 0024, Aachen
  - Local Institution - 0258, Berlin
  - Local Institution - 0020, Bonn
  - Local Institution - 0050, Cologne
  - Local Institution - 0026, Essen
  - Local Institution - 0093, Frankfurt am Main
  - Local Institution - 0040, Hanover
  - Local Institution - 0019, Homburg
  - Local Institution, Leipzig
  - Local Institution - 0036, Magdeburg
  - Local Institution - 0048, Mainz
  - Universitatsmedizin Mannheim, Mannheim
  - Local Institution - 0096, München
  - Local Institution - 0008, Tübingen
  - Local Institution, Würzburg
- Hong Kong (2):
  - Local Institution - 0120, Hong Kong
  - Local Institution - 0076, Hong Kong
- Italy (11):
  - Local Institution - 0136, Messina, ME
  - Local Institution - 0102, Bologna
  - Local Institution - 0077, Florence
  - Local Institution - 0104, Meldola
  - Local Institution - 0091, Milan
  - Local Institution, Modena
  - Local Institution - 0134, Monserrato
  - Local Institution - 0101, Napoli
  - Local Institution - 0119, Napoli
  - Local Institution - 0103, Padua
  - Local Institution - 0125, Rome
- Japan (21):
  - Local Institution - 0183, Kashiwa-shi, Chiba
  - Local Institution - 0201, Kurume-shi, Fukuoka
  - Local Institution - 0200, Sapporo, Hokkaido
  - Local Institution - 0184, Sapporo, Hokkaido
  - Local Institution - 0216, Nishinomiya-shi, Hyōgo
  - Local Institution - 0257, Morioka, Iwate
  - Local Institution - 0202, Kumamoto, Kumamoto
  - Local Institution - 0203, Osaka, Osaka
  - Local Institution - 0198, Osaka, Osaka
  - Local Institution, Ōsaka-sayama, Osaka
  - Local Institution - 0214, Suita-shi, Osaka
  - Local Institution - 0185, Tokushima, Tokushima
  - Local Institution - 0215, Bunkyo-ku, Tokyo
  - Local Institution - 0196, Chuo-ku, Tokyo
  - Local Institution - 0182, Mitaka-shi, Tokyo
  - Local Institution - 0210, Musashino-shi, Tokyo
  - Local Institution - 0186, Shinjuku-ku, Tokyo
  - Local Institution - 0187, Chiba
  - Local Institution - 0179, Hiroshima
  - Local Institution - 0180, Ishikawa
  - Local Institution - 0197, Kanagawa
- Mexico (4):
  - Local Institution - 0148, Cuauhtémoc, Durango
  - Local Institution - 0121, Monterrey, Nuevo León
  - Local Institution - 0264, Monterrey, Nuevo León
  - Local Institution - 0226, San Luis Potosí City
- Netherlands (2):
  - Local Institution - 0263, Maastricht
  - Local Institution - 0260, Utrecht
- Local Institution - 0240, Auckland, New Zealand
- Local Institution - 0231, San Juan, Puerto Rico
- Romania (6):
  - Local Institution, Brasov
  - Local Institution - 0078, Bucharest
  - Local Institution - 0232, Cluj-Napoca
  - Local Institution - 0242, Constanța
  - Local Institution - 0074, Craiova
  - Local Institution - 0070, Timișoara
- Russia (4):
  - Local Institution - 0032, Saint Petersburg, Sankt-Peterburg
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - Local Institution, Leningrad Region
  - Local Institution - 0230, Moscow
- Singapore (3):
  - Local Institution - 0042, Singapore
  - Local Institution - 0067, Singapore
  - Local Institution - 0039, Singapore
- South Korea (12):
  - Local Institution - 0191, Suwon, Gyeonggi-do
  - Local Institution - 0127, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0177, Daegu
  - Local Institution - 0190, Goyang-si
  - Local Institution - 0188, Gyeongsangnam-do
  - Local Institution - 0178, Jeollanam-do
  - Local Institution - 0169, Seongnam-si
  - Local Institution - 0128, Seoul
  - Local Institution - 0168, Seoul
  - Local Institution - 0167, Seoul
  - Local Institution - 0195, Seoul
  - Local Institution - 0189, Seoul
- Spain (11):
  - Local Institution - 0069, Barcelona
  - Local Institution - 0031, Barcelona
  - Local Institution - 0016, Córdoba
  - Local Institution - 0072, Donostia / San Sebastian
  - Local Institution - 0199, Madrid
  - Local Institution - 0109, Madrid
  - Local Institution - 0100, Pamplona
  - Local Institution - 0010, Sabadell (Barcelona)
  - Local Institution - 0028, Seville
  - Local Institution - 0082, Valencia
  - Local Institution - 0097, Zaragoza
- Taiwan (10):
  - Local Institution - 0131, Tainan, TNN
  - Local Institution - 0204, Kaohsiung City
  - Local Institution - 0130, Taichung
  - Local Institution - 0140, Taichung
  - Local Institution - 0174, Tainan
  - Local Institution - 0207, Taipei
  - Local Institution - 0173, Taipei
  - Local Institution - 0129, Taipei
  - Local Institution - 0175, Taoyuan District
  - Local Institution - 0176, Yunlin
- United Kingdom (5):
  - Local Institution - 0111, London
  - Local Institution - 0092, London
  - Local Institution - 0153, London
  - Local Institution - 0114, Manchester
  - Local Institution - 0142, Metropolitan Borough of Wirral

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03383458.html